CLINICAL TRIAL: NCT00755261
Title: Phase II Study of Doxorubicin and Avastin® for Patients With Advanced Soft-tissue Sarcomas.
Brief Title: Phase II Study of Doxorubicin and Avastin® in Sarcoma.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated due to low accrual.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J07133; NA_00013238 (Other: Johns Hopkins University IRB); AVF3855s (Other: Genentech, Inc)
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Sarcoma; Soft Tissue Sarcoma
Keywords: STS
MeSH Terms: conditions — Sarcoma | interventions — Bevacizumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin and Doxorubicin (Experimental): Patients will be treated with Avastin 15 mg/kg IV infusion plus doxorubicin 60 mg/M2 (body surface area) IV 6-hour infusion on Day 1 of each 21-day treatment cycle. Dose reductions/modifications will be applied as indicated by toxicities and/or patient tolerance.
  Interventions: Drug: Avastin; Drug: Doxorubicin

INTERVENTIONS:
Drug: Avastin — Combination of Avastin and doxorubicin. If initial 90 +/- 15 minute infusion of Avastin is tolerated without fever and chills, the 2nd dose may be infused over 60 +/- 10 minutes. If well tolerated, all subsequent infusions may be delivered over 30 +/- 10 minutes.
  Other Names: bevacizumab
Drug: Doxorubicin — The Day 1 6- hour continuous IV infusion must be done through a central venous catheter.
  Other Names: Adriamycin

SUMMARY:
This research is being done to find out if adding a drug called Avastin to an already approved regimen used for soft-tissue sarcoma, Doxorubicin, will improve overall survival, and slow disease progression. The study will also evaluate the overall safety of combining these drugs. It is not known if combining these drugs will improve outcome. Avastin has been approved for the treatment of metastatic carcinoma of the colon or rectum. It is not approved for the treatment of soft-tissue sarcoma when added to Doxorubicin.

DETAILED DESCRIPTION:
The rationale for this trial is to improve the efficacy of prototypical anti-sarcoma chemotherapeutic regimen Doxorubicin when combined with Avastin®. Soft tissue sarcomas are highly vascular tumors and are therefore ideally suited to trials combining angiogenic inhibitors with chemotherapy. Several studies have revealed correlations between prognosis and surrogates for angiogenesis, including microvessel density, and circulating VEGF and basic fibroblast growth factor (bFGF). The aim of this study is to evaluate the safety and efficacy of Avastin® in combination with Doxorubicin for the treatment of advanced soft-tissue sarcomas.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed intermediate or high grade locally advanced or metastatic soft tissue sarcoma.
2. The presence of measurable disease
3. Normal renal function (spot dipstick <2** or urine protein: creatinine ratio >1.0
4. Normal Hepatic function (total bilirubin within JOHC normal limits, transaminases (AST and ALT <3 times upper limit of normal
5. Hematologic parameters as defined as ANC >1500/mm³ and Platelets > 100,000/mm³.
6. Performance status 0-1 on ECOG scale
7. Use of effective means of contraception (men and women) in subjects of child-bearing age
8. No prior use of mesna, adriamycin, ifosfamide or Avastin®.
9. Baseline ECHO or MUGA with LVEF > or = 50-60%.
10. Age ≥ 18

Exclusion Criteria:

1. Major surgery within 28 days
2. History of proteinuria > 1+
3. Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored Avastin® cancer study
4. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
5. Any prior history of hypertensive crisis or hypertensive encephalopathy
6. New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
7. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
8. History of stroke or transient ischemic attack within 6 months prior to study enrollment
9. Symptomatic peripheral vascular disease
10. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
11. Evidence of bleeding diathesis or coagulopathy
12. Current or recent (within 10 days of enrollment) use of aspirin (>325 mg/day) or chronic use of other NSAIDs
13. Current, ongoing treatment with full-dose warfarin or its equivalent (i.e., unfractionated and/or low molecular weight heparin).
14. Known central nervous system or brain metastases
15. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
16. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
17. Pregnant (positive pregnancy test) or lactating
18. Proteinuria :creatinine (UPC) ratio ≥ 1.0 at screening or Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
19. History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
20. Serious, non-healing wound, ulcer, or bone fracture
21. Known hypersensitivity to any component of Avastin®
22. Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A Thornton, MD, Principal Investigator — Johns Hopkins SKCCC
Locations (1):
- Johns Hopkins SKCCC, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 4 subjects were accrued over 2 years. Study was closed due to slow accrual.
Period: Overall Study
Arm/Group | Avastin and Doxorubicin
Started | 6
Completed | 4
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Avastin and Doxorubicin
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 58 [45 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: RECIST
Description: Study was terminated because of low accrual.
Time Frame: 6 month PFS
Population: study was terminated because of low accrual (4 subjects enrolled/2 years)
Arm/Group | Avastin and Doxorubicin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: none, study was terminated early because of low accrual.
Arm/Group | Avastin and Doxorubicin
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin and Doxorubicin (N=4)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) — Oral thrush, dehydration, no able to swallow medications. No oral intake x 5 days.
acute renal failure (Renal and urinary disorders) | 1 (1) — Known pelvic malignancy; limited urinary sx. Scr creatinine = 0.9. Unable to void 24- 36 hrs. No output with straight catheterization. Creatinine=5.3. Occurred prior to any oral study drug being taken. Not related to treatment.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avastin and Doxorubicin (N=4)
thrush (Infections and infestations) | 1 (4)
dehydration (Metabolism and nutrition disorders) | 1 (1)
dysphagia -unable to swallow medications (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days